CLINICAL TRIAL: NCT01508793
Title: Enhancing Sleep Duration: Effects on Children's Eating and Activity Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL092910 (NIH)
Record Dates: First submitted 2012-01-05; First posted 2012-01-12 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Sleep; Obesity
Keywords: Sleep; Obesity; Children; Eating behaviors; Activity
MeSH Terms: conditions — Obesity; Feeding Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Optimize Sleep (Experimental)
  Interventions: Behavioral: Optimize Sleep

INTERVENTIONS:
Behavioral: Optimize Sleep — Children are asked to increase their sleep by approximately 1 1/2 hours/night for the duration of the two month intervention
  Arms: Optimize Sleep

SUMMARY:
The proposed study aims to determine whether an intervention to increase sleep in school-age children is associated with positive changes in eating, activity behaviors and zBMI. One hundred four children 8-11 years old who sleep 9 ½ hours or less per night will be randomly assigned to 1 of 2 conditions: 1) optimize sleep (increase TIB by 1 ½ hours/night to produce a change in sleep duration of approximately 40 minutes/night), or 2) control (no change in sleep). Families of children in the optimize sleep group will be taught effective behavioral strategies that have been shown to improve sleep duration. At baseline, 2-week and 2-month follow-up, the following will be gathered: sleep duration (measured by actigraphy), food intake (measured by 3 days of 24-hour recall), activity level (measured by accelerometry), the relative reinforcing value (RRV) of food (measured using a validated experimental paradigm), and measured child height and weight.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-11 years old
* BMI for age and gender > 10th percentile (but no greater than 100% overweight)
* Sleep 9.5 hours or less nightly
* Attend elementary school
* Like at least 1 food used in the reinforcement paradigm
* Able to understand and complete the reinforcement paradigm

Exclusion Criteria:

* Existence of a diagnosable parasomnia, sleep disordered breathing
* Medical or psychiatric condition that could influence sleep or weight
* Inability to complete study materials, including diagnosed disabilities
* Dietary restrictions/allergies to foods used in the study that preclude them from study participation

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Duration | Baseline, 2-weeks, and 2-months
  Measured with actigraphy
Change in Dietary Intake | Baseline, 2-weeks, and 2-months
  Measured using 24-hour dietary recalls (2 weekday and 1 weekend day)

SECONDARY OUTCOMES:
Change in the Reinforcing Value of Food | Baseline, 2-weeks, and 2-months
  Measured using a computer paradigm, the Behavioral Choice Task
Change in activity | Baseline, 2-week, and 2-month
  Physical and sedentary activities assessed using accelerometers and self-report
Change in zBMI | Baseline, 2-week, and 2-month
  Based on measured height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Chantelle N Hart, Ph.D., Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Center for Obesity Research and Education, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island